CLINICAL TRIAL: NCT03251339
Title: A Randomized, Double-blind, Parallel Group,Controlled Study to Compare the Immunogenicity and Safety of MSB11455 and Neulasta® in Healthy Adult Subjects
Brief Title: Safety and Immunogenicity of MSB11455 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fresenius Kabi SwissBioSim GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: EMR200621-003
Record Dates: First submitted 2017-08-15; First posted 2017-08-16 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-03

CONDITIONS: Healthy
Keywords: Healthy Participants; MSB11455
MeSH Terms: interventions — pegfilgrastim

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MSB11455 (Experimental): Participants received a single subcutaneous injection of MSB11455 6 milligram (mg) per (/) 0.6 milliliter (mL) on Day 1 in morning of treatment period 1 (28 Days) and 2 (28 Days). Period 1 and Period 2 are separated by a washout period of 35 Days.
  Interventions: Drug: MSB11455
- US-Neulasta (Experimental): Participants received a single subcutaneous injection of US-Neulasta 6 mg/0.6 mL on Day 1 in morning of treatment period 1 and 2. Period 1 and Period 2 are separated by a washout period of 35 Days.
  Interventions: Drug: US-Neulasta

INTERVENTIONS:
Drug: MSB11455 — Participants received a single subcutaneous injection of MSB11455 6 milligram (mg) per (/) 0.6 milliliter (mL) on Day 1 in morning of treatment period 1 (28 Days) and 2 (28 Days). Period 1 and Period 2 are separated by a washout period of 35 Days.
  Arms: MSB11455
Drug: US-Neulasta — Participants received a single subcutaneous injection of US-Neulasta 6 mg/0.6 mL on Day 1 in morning of treatment period 1 and 2. Period 1 and Period 2 are separated by a washout period of 35 Days.
  Other Names: pegfilgrastim
  Arms: US-Neulasta

SUMMARY:
The primary purpose of this study is to compare the immunogenicity and safety of MSB11455 and Neulasta in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants who provide signed and dated written informed consent.
* Participants with laboratory test results within predefined ranges.
* Other protocol defined inclusion criteria could apply.

Exclusion Criteria:

* Participants with known hypersensitivity to any component of US-Neulasta or MSB11455.
* Other protocol defined exclusion criteria could apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 336 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2018-02-05 (Actual); Study Completion 2018-09-22 (Actual)

PRIMARY OUTCOMES:
To Assess the Immunogenicity of MSB11455 Compared to Neulasta | From first dose up to end of study (Up to 3 months)
  Immunogenicity assessment will be based on Antidrug Antibody (ADA) response and development of Neutralizing Antibodies (NAB)

SECONDARY OUTCOMES:
Safety Profile as Assessed by Clinical Adverse events (AEs), Laboratory Variables, Vital Signs, Incidence of Antidrug Antibodies (ADAs), Neutralizing Antibodies(NABs) | Day 1 up to a maximum of 1 year
  Safety assessment will be based on number of subjects with AEs, abnormal laboratory variables, abnormal vital signs, incidence of ADAs and NABs

CONTACTS AND LOCATIONS:
Overall Officials: Radmila Kanceva, MD, PhD, Study Director — Fresenius Kabi SwissBioSim
Locations (2):
- New Zealand (2):
  - Auckland Clinical Studies Ltd, Auckland
  - Christchurch Clinical Studies Trust, Christchurch